CLINICAL TRIAL: NCT06672848
Title: Comparison of the Effects of Erector Spinae Area (ESP) Block and Thoracic Paravertebral Block (TPVB) on Acute Pain, Postoperative Persistent Pain and Neuropathic Pain in Video-Assisted Thoracoscopic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, MD, Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: E-53043469-050.04-613082
Record Dates: First submitted 2024-10-21; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
Keywords: postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomized double blinding
Who Masked: Participant, Care Provider
Masking Description: Blind patients and postoperative follow-ups will not know which group the patient is in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- esp block (Other): After anesthesia and surgical procedures, an ESP block will be applied under ultrasonography guidance from the midline 3 cm lateral from the T5 level. After cleaning the area with povidone-iodine before the block, the T5 transverse protrusion will be determined using a linear ultrasound probe. Local anesthetic will be applied between the transverse process and the erector spinae muscle with the help of an insulated needle designed for peripheral block procedures. The location of the needle will be confirmed by hydrodissection with physiological saline without local anesthesia. Once the location of the needle is confirmed, a mixture of 20 ml of 0.25% bupivacaine will be applied.
  Interventions: Diagnostic Test: Numeretic rating scale (NRS); Diagnostic Test: Brief Pain Inventory (BPI); Diagnostic Test: The S-LANSS Pain Score
- paravertebral block (Other): Following anesthesia and the surgical procedure, the needle will be advanced at an angle of 30-40° under ultrasonography guidance in the paramedian sagittal plane, lateral to the T5 spinos process, and entered into the location of the superior costotransverse ligament. The location of the serum and needle will be confirmed by hydrodissection without local anesthesia. Once the location of the needle is confirmed, a mixture of 20 ml of 0.25% bupivacaine will be applied.
  Interventions: Diagnostic Test: Numeretic rating scale (NRS); Diagnostic Test: Brief Pain Inventory (BPI); Diagnostic Test: The S-LANSS Pain Score

INTERVENTIONS:
Diagnostic Test: Numeretic rating scale (NRS) — NRS is a pain intensity determination system based on the person being asked to describe their pain on a scale of 0 (none), 10 (unbearable pain) and a point between.
Diagnostic Test: Brief Pain Inventory (BPI) — BPI is a chronic pain intensity determination system based on the person being asked to describe their pain on a scale of 0 (none), 10 (unbearable pain) and a point between.
Diagnostic Test: The S-LANSS Pain Score — The Leeds assessment of neuropathic symptoms and signs (LANSS) Pain Scale is based on analysis of sensory description and bedside examination of sensory dysfunction, and provides immediate information in clinical settings. It was developed in two populations of chronic pain patients.

SUMMARY:
VATS is a minimally invasive approach that allows the introduction of a video camera and surgical instruments into the thoracic cavity through small incisions made in the chest wall. The first thoracoscopy was performed by Jacobeus in 1910, and a cystoscope was used in this procedure. Over the years, with the development of surgical techniques and technology, the procedures performed using VATS have diversified. Today, it is used for the diagnosis of pleural diseases and effusions, the staging of lung cancer, lung lobectomies, and the determination of parenchymal diseases.

Respiratory therapy and pain management after extubation are important issues in postoperative care. Adequate postoperative pain control is necessary for a good respiratory effort. The use of intravenous opioids has become the standard in pain management for years. Opioids administered to adequately control pain can cause sedation and respiratory depression. Due to the large number of opioid-related side effects, alternative pain relief methods are being sought. Erector spinae area (ESP) block and thoracic paravertebral block (TPVB) have recently been described for the treatment of pain after thoracic surgery. Although these blocks have been shown to be effective in the treatment of pain after thoracotomy when compared with systemically administered opioids, they have not been compared in terms of the quality of recovery and postoperative pain after minimally invasive thoracic surgery.

The aim of this clinical trial is to compare the effects of Erector Spinae Area (ESP) Block and Thoracic Paravertebral Block (TPVB) on postoperative acute pain in patients scheduled for VATS surgery. The effects of the 2 blocks on postoperative chronic pain and neuropathic pain will also be compared.

Participants:

Their pain status will be recorded for 24 hours after spinal surgery When they come for a follow-up visit 3 months after surgery, 2 tests will be performed to check their pain status.

ELIGIBILITY:
Inclusion Criteria:

* Elective VATS surgery performed
* ASA I-III
* 18-75 years old

Exclusion Criteria:

* 1. Refusal at enrollment 2. Request for withdrawal from the study 3. Inability to give informed consent 4. Emergency surgery 5. Bleeding diathesis 6. Presence of contraindications to the LA agents used in this study 7. Use of chronic opioids 8. Psychiatric disorders 9. Presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
acute postoperative pain | Patients' pain levels and NRS scores will be recorded in the preoperative period and at the 1st, 6th, 12th, 24th and 48th hours postoperatively.
  NRS is a pain intensity determination system based on the person being asked to describe their pain on a scale of 0 (none), 10 (unbearable pain) and a point between

SECONDARY OUTCOMES:
chronic persistent pain and neuropatic pain | At the 3rd postoperative month, chronic persistent pain will be evaluated with BPI and neuropathic pain will be evaluated with the S-LANSS scoring system.
  BPI Scoring Patients are asked to rate their current symptoms, their average experiences of pain, and the minimum and maximum intensities of their symptoms on scales that range from 0 to 10. A total pain severity score can be found by averag- ing these items or a single item can be treated as the primary outcome measure. A score relating to impact on daily life can be calculated by averag- ing scores on each of the seven items, which also use scales from 0 to 10. Higher scores indicate greater severity and more interference.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fu Z, Zhang Y, Zhou Y, Li Z, Wang K, Li H, Jiang W, Liu Z, Cao X. A comparison of paravertebral block, erector spinae plane block and the combination of erector spinae plane block and paravertebral block for post-operative analgesia after video-assisted thoracoscopic surgery: A randomised controlled trial. J Minim Access Surg. 2022 Apr-Jun;18(2):241-247. doi: 10.4103/jmas.JMAS_277_20. PMID 33885016